CLINICAL TRIAL: NCT03589170
Title: Atrial Fibrilation Opportunistic Screening and Stroke Incidence (AFOSS): Searching the Unknown Atrial Fibrillation.
Brief Title: ATRIAL FIBRILATION OPPORTUNISTIC SCREENING AND STROKE (AFOSS).
Acronym: AFOSS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: University Rovira i Virgili (Other); Catalan Institute of Health (Other Government)
Responsible Party: Sponsor
Other Study IDs: 10-ECO
Record Dates: First submitted 2018-07-05; First posted 2018-07-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Opportunistic screening; ischaemic stroke
MeSH Terms: conditions — Atrial Fibrillation; Ischemic Stroke

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People over 60 years of age: People over 60 years of age without previous known atrial fibrillation
  Interventions: Diagnostic Test: Opportunistic atrial fibrillation screening

INTERVENTIONS:
Diagnostic Test: Opportunistic atrial fibrillation screening — Opportunistic pulse palpation and/or ECG at least once a year when they visit doctors or nurse for other reasons.
  Other Names: detection atrial fibrillation; pulse palpation

SUMMARY:
People: The absolute prevalence of undiagnosed atrial fibrillation in individuals over 60 years of age is 2.2%, equivalent to 20.1% of the overall prevalence of AF and there is not sufficient evidence regarding the procedures that may be most effective for achieving an early diagnosis of AF and reducing the associated stroke risks.

Intervention: Characterize the ideal population for searching unknown atrial fibrillation and develop an understanding of actions that could be taken today to improve the diagnosis and management of AF.

C: Compare two large populations with and without opportunistic screening of AF about stroke incidence.

Outcome: MAIN OBJECTIVES

1. Compare two large populations with and without opportunistic screening of AF.
2. Relate the incidence of stroke episode with the AF diagnosis
3. Characterize the ideal population for searching unknown atrial fibrillation by making a multivariate predictor model.
4. Develop an understanding of actions that could be taken today to improve the diagnosis and management of AF.
5. Evaluate whether intervention results in improved outcomes

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common arrhythmia encountered in clinical practice, and is increasing in both incidence and prevalence. Almost two hundred thousand Catalonian people over 60 year-old currently have AF, and estimates project that between 250.000 and 300.000 will be affected by 2050. Perhaps the most important consequence of AF is the risk of embolic stroke.

It has been estimated that around one in five strokes are attributed to AF overall, and one in three strokes in people over the age of 80 are attributed to AF. AF-related strokes are associated with significant morbidity, mortality and healthcare costs, yet they are highly preventable. Unfortunately, AF is often undiagnosed or untreated when stroke occurs.

In addition, the absolute prevalence of undiagnosed atrial fibrillation in individuals over 60 years of age is 2.2%, equivalent to 20.1% of the overall prevalence of AF. This is higher than in the reports of other studies, which range from 0.49% to 1.7% when diagnosed by means of standard ECG, but lower than the AF incidence (30%) detected by continuous monitoring in patients with risk factors for stroke. The prevalence of AF in the community is probably underestimated, as a consequence of the failure to detect and diagnose it and may be responsible for an additional subset of the 25-40% of strokes of unknown cause. It has been suggested that asymptomatic AF represents a third of the total AF population, a result confirmed in pacemaker studies. Around thirty eight thousand Catalonian people over 60 year-old currently could suffer unknown AF, and consequently non-treated, and estimates project that between 1,350-2,475 stroke/year could be related to this untreated condition.

While the data confirm the evident age-related increase in the prevalence of persistent AF and demonstrate that hypertension is the most frequently associated cardiovascular risk factor together with the presence of cardiovascular disease there is not sufficient evidence regarding the procedures that may be most effective for achieving an early diagnosis of AF and reducing the associated risks. A significant proportion of people with AF are diag¬nosed by chance during health assessments carried out for other reasons, or due to having a stroke. There may be multiple reasons for under-diagnosis, including the fact that AF can be asymptomatic and a lack of awareness about the condition and its symptoms. There is considerable interest in developing AF screening programs

Opportunistic screening, where patients are checked for AF when they visit doctors for other reasons, is widely supported as a means to achieve higher rates of detec¬tion to enable early intervention. Screening for AF anyone >65 years or at high risk of stroke has been recommended by Mention of European Society of Cardiology (ESC), Stroke Alliance for Europe (SAFE), European Heart Rhythm Association (EHRA), Royal College of Physicians of Edinburg (RCPE), World Healthcare Forum (WHF), European Primary Care Cardiovascular Society (EPCCS), Health Information and Quality Authority (HIQA), and AF-SCREEN. Currently, routine mass screenings are not carried out in any countries at a national level. Opportunistic screening was tested against routine screening by the SAFE study, which found that opportunistic screening improved on routine practice and out¬reach campaign in Spain[23] was found to have had little effect on diagnosis of previously undetected AF and it was concluded that opportunistic screening is thus a better strategy for early detection.

It is important to note that, for many patients with AF, the condition is often asymptomatic - or associated with minor symptoms that are ignored or unrecognized by patients - and some type of AF screening is needed. Until the new external devices can be used more widely, ECG combined with reviews of medical history will continue to be the most feasible noninvasive strategy for identifying individuals with AF in epidemiological studies. The key issue, however, is not which test is best for diagnosing AF or how to undertake an effective screening procedure, but it is rather the appropriate measurement of results and achieving optimal effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 60 years included in the computer program of the ICS (Catalan Institute of Health).

Exclusion Criteria:

* Patients under 60 years old. Deceased

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients over 60 years of age who have a medical history in the ICS (Catalan Institute of Health) in the Terres de l'Ebre region, Tarragona, Spain.
Sampling Method: Non-Probability Sample
Enrollment: 51410 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation | 01/Jan/2016 to 31/Decemb/2017
  Atrial fibrillation new diagnosis

SECONDARY OUTCOMES:
ischaemic stroke | 01/jan/2016 to 31/Decemb/2018
  New ischaemic stroke

CONTACTS AND LOCATIONS:
Overall Officials: Jose Maria Alegret-Colomè, PhD, Study Director — University Rovira i Virgili

IPD SHARING:
Plan to Share IPD: Yes
We will share information about our study at the end of the study if if they are valued positively.
Supporting Information: Study Protocol, CSR
Time Frame: At the end of the study.
Access Criteria: Applications received to share results will be independently assessed at the end of the study .

REFERENCES:
- [Result] Panisello-Tafalla A, Clua-Espuny JL, Gil-Guillen VF, Gonzalez-Henares A, Queralt-Tomas ML, Lopez-Pablo C, Lucas-Noll J, Lechuga-Duran I, Ripolles-Vicente R, Carot-Domenech J, Lopez MG. Results from the Registry of Atrial Fibrillation (AFABE): Gap between Undiagnosed and Registered Atrial Fibrillation in Adults--Ineffectiveness of Oral Anticoagulation Treatment with VKA. Biomed Res Int. 2015;2015:134756. doi: 10.1155/2015/134756. Epub 2015 Jul 1. PMID 26229954
- [Result] Clua-Espuny JL, Lechuga-Duran I, Bosch-Princep R, Roso-Llorach A, Panisello-Tafalla A, Lucas-Noll J, Lopez-Pablo C, Queralt-Tomas L, Gimenez-Garcia E, Gonzalez-Rojas N, Gallofre Lopez M. Prevalence of undiagnosed atrial fibrillation and of that not being treated with anticoagulant drugs: the AFABE study. Rev Esp Cardiol (Engl Ed). 2013 Jul;66(7):545-52. doi: 10.1016/j.rec.2013.03.003. Epub 2013 May 31. PMID 24776203
- [Result] Clua-Espuny JL, Panisello-Tafalla A, Lopez-Pablo C, Lechuga-Duran I, Bosch-Princep R, Lucas-Noll J, Gonzalez-Henares A, Queralt-Tomas L, Ripolles-Vicente R, Calduch-Noll C, Gonzalez-Rojas N, Gallofre-Lopez M. Atrial Fibrillation and Cardiovascular Comorbidities, Survival and Mortality: A Real-Life Observational Study. Cardiol Res. 2014 Feb;5(1):12-22. doi: 10.14740/cr324e. Epub 2014 Feb 27. PMID 28392870
- [Result] Clua-Espuny JL, Pinol-Moreso JL, Gil-Guillen VF, Orozco-Beltran D, Panisello-Tafalla A, Lucas-Noll J, Queralt-Tomas ML, Pla-Farnos R. [Primary and secondary cardiovascular prevention results in patients with stroke: relapse risk and associated survival (Ebrictus study)]. Rev Neurol. 2012 Jan 16;54(2):81-92. Spanish. PMID 22234566
- [Result] Clua Espuny JL, Dalmau Llorca MR, Aguilar Martin C; Grupo de Trabajo. [Characteristics of oral anti-coagulation treatment in high-risk chronic auricular fibrillation]. Aten Primaria. 2004 Nov 15;34(8):414-9. doi: 10.1016/s0212-6567(04)78925-8. Spanish. PMID 15546539
- [Result] Gimenez-Garcia E, Clua-Espuny JL, Bosch-Princep R, Lopez-Pablo C, Lechuga-Duran I, Gallofre-Lopez M, Panisello-Tafalla A, Lucas-Noll J, Queralt-Tomas ML. [The management of atrial fibrillation and characteristics of its current care in outpatients. AFABE observational study]. Aten Primaria. 2014 Feb;46(2):58-67. doi: 10.1016/j.aprim.2013.06.003. Epub 2013 Sep 14. Spanish. PMID 24042075